CLINICAL TRIAL: NCT06300918
Title: A Randomized Controlled Clinical Trial to Evaluate the Time Point of Anti-VEGF Pretreatment of PDR Based on Intraoperative FFA
Brief Title: A Clinical Trial to Evaluate the Time Point of Anti-VEGF Pretreatment of PDR Based on Intraoperative FFA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jie Li (Other)
Responsible Party: Sponsor-Investigator, Jie Li, Principal Investigator, Sichuan Provincial People's Hospital
Organization: Sichuan Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2024-KY76
Record Dates: First submitted 2024-02-22; First posted 2024-03-08 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: The Condition of Fundus Neovascularization
MeSH Terms: interventions — Time

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Injecting anti-VEGF drugs 3 days before operation (Experimental): Injecting Conbercept into vitreous cavity 3 days before performing vitrectomy.
  Interventions: Other: Time
- Injecting anti-VEGF drugs 7 days before operation (Experimental): Injecting Conbercept into vitreous cavity 7 days before performing vitrectomy.
  Interventions: Other: Time
- Injecting anti-VEGF drugs 14 days before operation (Experimental): Injecting Conbercept into vitreous cavity 14 days before performing vitrectomy.
  Interventions: Other: Time

INTERVENTIONS:
Other: Time — Time point of injecting anti-VEGF drugs

SUMMARY:
The goal of this prospective randomized controlled study is to compare the therapeutic effect of injecting anti-VEGF drugs before surgery for patients with proliferative diabetic retinopathy at different time points. At present, studies have confirmed that anti-VEGF drugs are effective in inhibiting fundus neovascularization in proliferative diabetic retinopathy. The main question it aims to answer is which time point is better to injecting anti-VEGF drugs before surgery for patients with proliferative diabetic retinopathy.

Participants will be randomly divided into three groups. And time points of injecting anti-VEGF drugs before surgery for each group will be 3 days, 7 days, 14 days. And we have a new technology that can have fluorescein fundus angiography during operation, so it can reflect the condition of fundus neovascularization immediately and precisely. In that case, we can compare the Inhibitory effect of anti-VEGF drugs on fundus neovascularization at different time points.

ELIGIBILITY:
Inclusion Criteria:

* PDR is diagnosed in people 18 years of age or older with type 1 or type 2 diabetes，
* Hemoglobin A1c (HbA1c) ≤10%
* Persistent vitreous hemorrhage for more than one month or recurrent vitreous hemorrhage (within six months)
* Did not undergo retintis photocoagulation (PRP)
* Vitreous hemorrhage disease course within six months

Exclusion Criteria:

* Patients who have had previous vitreoretinal surgery
* Intravitreal drug injection within 3 months
* Eye diseases other than PDR that may hinder vision improvement, such as optic atrophy or macular hole
* Thromboembolic events (including cerebrovascular or myocardial infarction) or clotting system disorders or receiving anticoagulation or antiplatelet therapy
* B-ultrasound or indirect fundus microscopy showing retina detachment (pull or hole origin)
* Vitrectomy, FFA contraindicated patients, patients with severe abnormality of cardiopulmonary, liver and kidney function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
The number of fundus neovascularization seen in FFA. | Observed during operation
  Fundus neovascularization
The area of fundus neovascularization seen in FFA (using PD size as measurement). | Observed during operation
  Fundus neovascularization
The intensity of neovascularization fluorescein leakage | Observed during operation
  2- and 5-minute images were taken to assess the intensity of neovascularization fluorescein leakage through FFA.Fluorescein leakage intensity classification and leakage score (judged by postoperative video or jigsaw puzzle) : no leakage is 0; The suspected leakage was level 1. It is clear that the expansion range of leakage point is less than 1PD, which is grade 2. It is clear that leakage greater than or equal to 1PD is grade 3; Leakage integral is the sum of leakage number x leakage strength classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Academy of Medical Science Sichuan Provincial Hosptial, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
2030, via https://pan.baidu.com
Supporting Information: CSR
Time Frame: 2025 and forever
Access Criteria: via https://pan.baidu.com
URL: http://pan.baidu.com